# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT03548987 |
| Sponsor trial ID: | NN9536-4376 |
| Official title of study: | Effect and safety of semaglutide 2.4 mg once-weekly in subjects with overweight or obesity who have reached target dose during run-in period |
| Document date: | 25-June-2020 |

Semaglutide s.c. 2.4 mg once weekly Trial ID: NN9536-4376 (STEP 4) Clinical Trial Report Appendix 16.1.9


Date: Version: Status:

25 June 2020 | Novo Nordisk Final

## 16.1.9 Documentation of statistical methods

# List of contents

| Statistical analysis plan | Link |
|---------------------------|------|
| MedDRA searches | Link |

Redacted statistical analysis plan Includes redaction of personal identifiable information only.


Date: Version: Status: Page:

31 March 2020 Novo Nordisk 1.0 Final 1 of 24

# Statistical Analysis Plan

**Trial ID: NN9536-4376** 

# STEP 4

Effect and safety of semaglutide 2.4 mg once-weekly in subjects with overweight or obesity who have reached target dose during run-in period

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.


31 March 2020 | Novo Nordisk 1.0 Final 2 of 24

# **Table of contents**

| Tal | ole of co | tents | .2 |
|---|---|---|---|
| Lis | t of abb | eviations | .3 |
| 1 | Introd | ction | .5 |
| | 1.1 | Trial information | .5 |
| | | 1.1.1 Objective(s) | .5 |
| | | 1.1.1.1 Primary objective | .5 |
| | | 1.1.1.2 Secondary objectives | .5 |
| | | 1.1.2 Estimands | .5 |
| | 1.1.3 Endpoints | | |
| | | 1.1.3.1 Primary endpoint | .6 |
| | | 1.1.3.2 Secondary endpoints | .7 |
| | | 1.1.4 Type of trial | |
| | 1.2 | Scope of the statistical analysis plan | .8 |
| 2 | Statisti | al considerations | .9 |
| | 2.1 | Sample size determination | |
| | 2.2 | Definition of analysis sets1 | |
| | 2.3 | Statistical analyses | |
| | | 2.3.1 Primary endpoint | 2 |
| | | 2.3.2 Secondary endpoints1 | 7 |
| | | 2.3.2.1 Confirmatory secondary endpoints | 7 |
| | | 2.3.2.2 Supportive secondary endpoints | 8 |
| | | 2.3.3 Exploratory endpoints | 22 |
| | | 2.3.4 Other analyses | |
| | 2.4 | Pharmacokinetic and/or pharmacodynamic modelling | :2 |
| 3 | Change | s to the statistical analyses planned in the protocol2 | 23 |
| | 3.1 | Trial specific changes2 | |
| | 3.2 | Changes applied across STEP trials | |
| 4 | Refere | ces | 24 |

Statistical Analysis Plan Date: 31 March 2020 Novo Nordisk

 Trial ID: NN9536-4376
 Version:
 1.0

 UTN: U1111-1201-0898
 Status:
 Final

 EudraCT No.: 2017-003473-34
 Page:

## List of abbreviations

AD available but discontinued ANCOVA analysis of covariance

AT available on randomised treatment

BMI body mass index
BP bodily pain

CI confidence interval
dBP diastolic blood pressure
ECG electrocardiogram
FAS full analysis set
FFA free fatty acid

FPG fasting plasma glucose

GH general health

HbA1c glycated haemoglobin
HDL high density lipoprotein

*LAO-OT* last available observation during the on-treatment period

LDLlow-density lipoproteinMCSmental component summaryMDmissing and discontinued

MedDRA Medical Dictionary for Regulatory Activities

MH mental health

MMRM mixed model for repeated measurements

MT missing on randomised treatment PCS physical component summary

PF physical functioning
PYE patient years of exposure
PYO patient years of observation

RE role-emotional RP role-physical

SAE serious adverse event
SAP statistical analysis plan
SAS safety analysis set
sBP systolic blood pressure

s.c. subcutaneus

SD standard deviation SF social functioning SF-36 Short Form-36

TEAE treatment-emergent adverse event VLDL very low density lipoprotein


31 March 2020 | Novo Nordisk 1.0 Final 4 of 24

VTvitality

WCwaist circumference

WRSSM Weight Related Sign and Symptom Measure


31 March 2020 | Novo Nordisk 1.0 Final 5 of 24

#### Introduction 1

#### 1.1 **Trial information**

#### 1.1.1 Objective(s)

#### 1.1.1.1 Primary objective

Effect-related: randomisation (week 20) to week 68

To compare the effect of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as an adjunct to reduced-calorie diet and increased physical activity in subjects with overweight or obesity who have reached target dose of semaglutide during the run-in period, on body weight.

#### 1.1.1.2 Secondary objectives

Effect-related: randomisation (week 20) to week 68

To compare the effect of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as an adjunct to reduced-calorie diet and increased physical activity in subjects with overweight or obesity who have reached target dose of semaglutide during the run-in period, on

- cardiovascular risk factors
- clinical outcome assessments •
- glucose metabolism

Effect-related: week 0 to week 68

To investigate the effect of semaglutide s.c. 2.4 mg once-weekly as an adjunct to reduced-calorie diet and increased physical activity in subjects with overweight or obesity who have reached target dose during the run-in period, on body weight.

*Safety and tolerability: week 0 to randomisation (week 20)* 

To investigate the safety and tolerability of semaglutide s.c. 2.4 mg once-weekly as an adjunct to reduced-calorie diet and increased physical activity in subjects with overweight or obesity during the run-in period.

Safety and tolerability: randomisation (week 20) to week 75

To compare the safety and tolerability of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as an adjunct to reduced-calorie diet and increased physical activity in subjects with overweight or obesity who have reached target dose of semaglutide during the run-in period.

#### 1.1.2 **Estimands**

#### **Primary estimand**

The estimand will quantify the average treatment effect of semaglutide relative to semaglutide placebo after 48 weeks' treatment with semaglutide at the target dose, as an adjunct to reducedcalorie diet and increased physical activity, in all randomised subjects regardless of adherence to


31 March 2020 | Novo Nordisk 1.0 Final 6 of 24

treatment provided that the subjects are able to reach the target dose of semaglutide during 20 weeks run-in with escalating semaglutide doses and regardless of initiation of other anti-obesity therapies (i.e. weight management drugs or bariatric surgery) ("treatment policy" estimand).

The primary estimand will cover all effect-related objectives except the secondary objective addressing 'Effect-related: week 0 to week 68'.

### Secondary estimand

The estimand will quantify the average treatment effect of semaglutide relative to semaglutide placebo after 48 weeks' treatment with semaglutide at the target dose, as an adjunct to reducedcalorie diet and increased physical activity, in all randomised subjects had they remained on their randomised treatment for the entire 48 weeks after reaching the target dose of semaglutide during the 20 weeks run-in with escalating semaglutide doses and not initiated other anti-obesity therapies (i.e. weight management drugs or bariatric surgery) ("hypothetical" estimand).

The secondary estimand will cover all effect-related objectives except the secondary objective addressing 'Effect-related: week 0 to week 68'.

### **Tertiary estimand**

The estimand will quantify the average treatment effect of semaglutide after 68 weeks, as an adjunct to reduced-calorie diet and increased physical activity, in all randomised subjects regardless of adherence to treatment and regardless of initiation of other anti-obesity therapies (i.e. weight management drugs or bariatric surgery) ("treatment policy" estimand).

The tertiary estimand will cover the secondary objective addressing 'Effect-related: week 0 to week 68'.

### Quarternary estimand

The estimand will quantify the average treatment effect of semaglutide after 68 weeks, as an adjunct to reduced-calorie diet and increased physical activity, in all randomised subjects had they remained on their randomised treatment for the entire 68 weeks and not initiated other anti-obesity therapies (i.e. weight management drugs or bariatric surgery) ("hypothetical" estimand).

The quarternary estimand will cover the secondary objective addressing 'Effect-related: week 0 to week 68'.

#### 1.1.3 **Endpoints**

#### 1.1.3.1 **Primary endpoint**

Change from randomisation (week 20) to week 68 in body weight (%)

#### **CONFIDENTIAL**


31 March 2020 | Novo Nordisk 1.0 Final 7 of 24

#### 1.1.3.2 **Secondary endpoints**

### Confirmatory secondary endpoints

Effect endpoints from randomisation (week 20) to week 68 Change in:

- Waist circumference (cm)
- Systolic blood pressure (mmHg)
- Physical functioning score (SF-36)

### Supportive secondary endpoints

Effect endpoints from randomisation (week 20) to week 68 Change in:

- Body weight (kg)
- BMI  $(kg/m^2)$
- Haemoglobin A1c (HbA1c) (%, mmol/mol)
- Fasting plasma glucose (FPG) (mg/dL)
- Fasting serum insulin (mIU/L)
- Diastolic blood pressure (mmHg)
- Lipids (mg/dL)
  - o Total cholesterol
  - o High-density lipoproteins (HDL)
  - o Low-density lipoproteins (LDL)
  - Very low-density lipoproteins (VLDL)
  - o Free fatty acids
  - o Triglycerides
- SF-36:
- o Role-Physical score
- **Bodily Pain score**
- General Health score
- Vitality score
- Social Functioning score
- o Role-Emotional score
- Mental Health score
- Physical component summary
- Mental component summary

Subjects who achieve (yes/no):

Responder definition value for SF-36 physical functioning score

Subjects who gain weight (yes/no)


31 March 2020 | Novo Nordisk 1.0 Final 8 of 24

Effect endpoints from week 0 to week 68

Change in body weight (%)

Subjects who achieve (yes/no):

- Body weight reduction < 0%
- Body weight reduction  $\geq 5\%$
- Body weight reduction  $\geq 10\%$
- Body weight reduction  $\geq 15\%$
- Body weight reduction  $\geq 20\%$

Safety endpoints from week 0 to randomisation (week 20)

Number of treatment-emergent AEs

Number of serious adverse events (SAEs)

Change in:

- Pulse (bpm)
- Amylase (U/L)
- Lipase (U/L)
- Calcitonin (ng/L)

Safety endpoints from randomisation (week 20) to week 75 Number of treatment-emergent AEs Number of SAEs

Safety endpoints from randomisation (week 20) to week 68 Change in:

- Pulse (bpm)
- Amylase (U/L)
- Lipase (U/L)
- Calcitonin (ng/L)

#### 1.1.4 Type of trial

This is a 68-week, randomised, double-blind, placebo-controlled, two-armed multi-centre, multinational withdrawal clinical trial comparing once-weekly semaglutide s.c. 2.4 mg with semaglutide placebo in subjects with overweight or obesity.

#### 1.2 Scope of the statistical analysis plan

This statistical analysis plan (SAP) is based on the updated protocol for trial NN9536-4376 "Effect and safety of semaglutide 2.4 mg once-weekly in subjects with overweight or obesity who have reached target dose during run-in period", version 4.0 (04 September 2019) including amendment no. 3 (global), and includes more detailed procedures for executing the statistical analyses of the primary and secondary endpoints. Statistical analyses and a number of clarifications additional to

| Statistical Analysis Plan | Date: | 31 March 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: 2017-003473-34 | Page: | 9 of 24 | |

those specified in the trial protocol are pre-specified with this SAP. All changes to the statistical analyses planned in the trial protocol are documented in section  $\underline{3}$ .

### 2 Statistical considerations

### Taxonomy of week 68 assessments

For each subject a given assessment at week 68 may be available or missing and <u>Table 2-1</u> describes the taxonomy for this. Note, this is done per assessment and per subject; subjects may be a different type for different assessments (a subject may have "available on randomised treatment (AT)" for body weight but "missing on randomised treatment (MT)" for waist circumference).

Table 2-1 Taxonomy for subjects based on week 68 assessments

| Assessment<br>at week 68 | Subjects on<br>randomised<br>treatment at<br>week 68 | Type description | Type<br>Abbreviation |
|---|---|---|---|
| Available | Yes | Available on randomised treatment: Subjects who complete the trial on randomised treatment with an assessment at week 68: Includes those that stop and restart trial product | AT |
| | No | Available but discontinued Subjects who discontinued randomised treatment prematurely but returned to have an assessment at week 68. These are also called retrieved subjects | AD |
| Missing | Yes | Missing on randomised treatment: Subjects who complete the trial on randomised treatment without an assessment at week 68: Includes those that stop and restart trial product | MT |
| | No | Missing and discontinued: Subjects who discontinued randomised treatment prematurely and did not return to have an assessment at week 68. These are also called non-retrieved subjects | MD |

# 2.1 Sample size determination

The sample size and thereby the power for this trial is primarily defined to support safety. However, no formal statistical inference is planned based on number of adverse events. Given the trial sample size, the power of statistical tests for effect endpoints is described below.

The tests of superiority of semaglutide 2.4 mg to semaglutide placebo for the primary and confirmatory secondary endpoints are performed using the fixed-sequence statistical strategy. This strategy tests the endpoints using a predefined hierarchical order, all at the significance level of 5%, moving to test the next endpoint only after a statistically significant superiority result (p-value < 5%) on the previous endpoint. The test hierarchy is given in <u>Table 2-2</u> with underlying assumptions, marginal power and effective power. The effective power is calculated under the assumption of independence of endpoints by multiplying the respective marginal powers successively.

In the analysis approach addressing the primary estimand, week 68 assessments from retrieved subjects (AD) are used. These data are also used to impute missing measurements at week 68 for

 Statistical Analysis Plan
 Date:
 31 March 2020
 Novo Nordisk

 Trial ID: NN9536-4376
 Version:
 1.0
 1.0
 Status:
 Final
 Final
 Page:
 10 of 24</td

non-retrieved subjects (MD). The imputation is done separately within each treatment arm (see description below). However, for the power calculations missing values (MT and MD), regardless of treatment arm, are assumed to be similar to semaglutide placebo subjects. These assumptions are likely conservative with respect to the power, and correspond to the jump to reference sensitivity analysis planned below.

### **Assumptions**

The common assumptions for the power calculations are

- The significance level is 5%
- The randomisation ratio is 2:1
- For continuous endpoints the t-test on the mean difference assuming equal variances is used
- Based on data from NN9536-4153
  - 5% of subjects discontinue permanently between randomisation (week 20) and week
     68 and
  - o 60% of these are retrieved (AD) at week 68
- All subjects in the semaglutide placebo arm are assumed to have same effect as subjects who complete the trial on semaglutide placebo (AT)
- Retrieved subjects (AD) in the semaglutide 2.4 mg arm are assumed to have an effect
  corresponding to half the treatment difference (compared to semaglutide placebo) of
  subjects who complete the trial on semaglutide 2.4 mg (AT)
- Non-retrieved subjects (MD) in the semaglutide 2.4 mg arm are assumed to have an effect corresponding to semaglutide placebo

Further assumptions made to calculate the power for each of the primary and confirmatory secondary endpoints are based on findings from other projects conducted by Novo Nordisk (NN8022 (SCALE), NN9535 (SUSTAIN), NN9924 (PIONEER)), and trial NN9536-4153 and are presented in <u>Table 2-2</u>.

Given these assumptions, the sample size of 750 subjects (500 in the semaglutide 2.4 mg once weekly and 250 in the semaglutide placebo arm), gives an effective power (marginal powers multiplied) of 95% for the four endpoints in the hierarchical testing procedure. Under the additional assumption that minimum 80% of subjects will be eligible for randomisation a total of 900 subjects will be started on trial product. As sample size is primarily driven by safety, additional scenarios for assumptions are not included due to the overall high power.

| Statistical Analysis Plan | Date: | 31 March 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: 2017-003473-34 | Page: | 11 of 24 | |

Table 2-2 Assumptions, marginal power and effective power for each endpoint in the hierarchical testing procedure given an anticipated number of 750 randomised subjects

| Order | Endpoint | Assumed mean (±SD) for completers Semaglutide Semaglutide 2.4 mg placebo | | Expected mean<br>(±SD)<br>Semaglutide<br>2.4 mg | Expected<br>difference | Marginal<br>power<br>(%) | Effective power (%) |
|---|---|---|---|---|---|---|---|
| 1 | % weight change | -4 (±10) | +5 (±10) | -3.7 (±11) | 8.7 %-points | > 99 | > 99 |
| 2 | WC change (cm) | -3 (±10) | +3 (±10) | -2.8 (±11) | 5.8 cm | > 99 | > 99 |
| 3 | sBP change (mmHg) | -3.1 (±13) | +1 (±13) | -3 (±14) | 4 mmHg | 95 | 95 |
| 4 | SF-36 PF score change | +6 (±10) | +2 (±10) | +5.9 (±11) | 3.9 score-<br>points | > 99 | 95 |

SD = standard deviation; WC = waist circumference; sBP = systolic blood pressure; SF-36 = Short Form 36 v2.0 acute; PF = physical functioning

All tests in the hierarchy are based on the primary estimand

# 2.2 Definition of analysis sets

Two analysis sets are defined:

- The *full analysis set* (FAS) includes all randomised subjects according to the intention-to-treat principle. Subjects in the FAS will contribute to evaluation "as randomised".
- The *safety analysis set* (SAS) includes all subjects exposed to at least one dose of trial product. Subjects in the SAS will contribute to evaluation "as treated".

Any observation excluded from the analysis will be documented before database lock with the reason for exclusion provided.

Two observation periods are defined for each subject:

- In-trial: The *in-trial period* is defined as the uninterrupted time interval from date of week 0 to date of last contact with trial site.
- On-treatment (with trial product): A time-point is considered as 'on-treatment' if any dose of trial product has been administered within the prior 2 weeks (14 days). The *on-treatment period* is defined as all times which are considered on-treatment.
  - In general, the on-treatment period will therefore be from the date of first trial product administration to date of last trial product administration (+14 days) excluding potential off-treatment time intervals triggered by at least two consecutive missed doses.
  - For the evaluation of adverse events the lag time for each on-treatment time interval is 7 weeks (49 days) applicable to all subjects treated with trial product including those who are not eligible for randomisation.

The in-trial and on-treatment periods define the patient years of observation (PYO) and patient years of exposure (PYE), respectively, as the total time duration in the periods.


31 March 2020 | Novo Nordisk 1.0 Final 12 of 24

#### 2.3 Statistical analyses

If necessary, a statistical analysis plan (SAP) may be written in addition to the protocol, including a more technical and detailed elaboration of the statistical analyses. The SAP will be finalised before database lock.

Effect endpoints will be analysed using the FAS; safety endpoints will be analysed using the SAS.

Results from statistical analyses will generally be accompanied by two-sided 95% confidence intervals and corresponding p-values. Superiority will be claimed if p-values are less than 5% and the estimated treatment contrasts favours semaglutide 2.4 mg.

### Handling of missing baseline data

The last available and eligible observation at or before randomisation is used as the baseline (randomisation) value. If no assessments are available during the run-in period, the mean of baseline (randomisation) values across all subjects is used as the baseline (randomisation) value. For endpoints evaluating the change from week 0, the last available and eligible observation at or before the week 0 visit is used as the baseline (week 0) value. If no assessments are available, the mean of baseline (week 0) values across all subjects is used as the baseline (week 0) value.

#### 2.3.1 **Primary endpoint**

Definition of primary endpoint: % weight change

Change from baseline (randomisation/week 20) to week 68 in body weight (%) is defined as

% weight change = 
$$\frac{\text{(body weight at week 68 - body weight at baseline)}}{\text{body weight at baseline}} \times 100.$$

## Analyses addressing the primary estimand

The following statistical analysis and imputation methods are designed to address the primary estimand, i.e. to assess the effectiveness of semaglutide 2.4 mg.

The analysis model for % weight change is a linear regression (ANCOVA) of % weight change with randomised treatment as a factor and baseline body weight (kg) as covariate. The estimated treatment difference between semaglutide 2.4 mg and semaglutide placebo will be reported together with the associated two-sided 95% confidence interval (CI) and corresponding p-value.

The superiority tests of semaglutide 2.4 mg vs. semaglutide placebo will be carried out as follows.

Let  $\mu_{\text{semaglutide}}$  and  $\mu_{\text{semaglutide placebo}}$  denote the true mean of % weight change for semaglutide 2.4 mg and semaglutide placebo group, respectively. The null and alternative hypotheses tested are


31 March 2020 | Novo Nordisk 1.0 Final 13 of 24

 $H: \mu_{semaglutide} \geq \mu_{semaglutide\ placebo}\ vs$  $H_A$ :  $\mu_{semaglutide} < \mu_{semaglutide\ placebo}$ .

The hypothesis will be rejected and superiority claimed, if the upper limit of the estimated twosided 95% CI is below 0.

Handling of missing week 68 values for the primary estimand

All available data at week 68 (AT and AD) are used and missing values (MT and MD) at week 68 will be imputed and the endpoint will be derived from the imputed values. Several approaches for imputation will be applied. First, a description of the primary imputation approach to address the primary estimand for the primary endpoint is given followed by a description of the sensitivity analyses used to assess the robustness of the primary analysis results. The sensitivity analyses investigate how assumptions on body weight development after discontinuation of randomised treatment impact the estimated treatment contrasts between semaglutide 2.4 mg and semaglutide placebo. An illustration of all imputation approaches for the primary estimand is given in Figure 2-1.

Primary imputation approach for the primary estimand

Multiple imputation approach using retrieved subjects (RD-MI): The primary imputation approach for the primary estimand is a multiple imputation similar to the one described by McEvoy.<sup>2</sup> Missing body weight measurement at week 68 for non-retrieved subjects (MD) are imputed using assessments from retrieved subjects (AD) in each randomised treatment arm. This will be done according to the timing of last available observation on-treatment (LAO-OT) of body weight prior to week 68. Missing body weight measurements at week 68 for subjects on randomised treatment (MT) are imputed in a similar way by sampling from available measurements at week 68 from subjects on randomised treatment (AT) in the relevant randomised treatment arm. The multiple imputation approach is done in three steps:

1. **Imputation**: Defines an imputation model using retrieved subjects (AD) from FAS and done within groups defined by randomised treatment. The model will be a linear regression of body weight (kg) at week 68 with gender (male/female), baseline BMI (kg/m<sup>2</sup>) (in categories  $\leq$ 35, 35-<40, ≥40) and timing of the LAO-OT of body weight as factors and baseline (randomisation) body weight (kg) and LAO-OT of body weight (kg) as covariates. No interactions will be included. The grouping of timing will be done by quarters (intervals of 12 weeks for endpoints evaluating the change from randomisation, intervals of 17 weeks for endpoints evaluating the change from week 0). If timing by quarters is too restrictive, halves (intervals of 24 weeks for endpoints evaluating the change from randomisation, intervals of 34 weeks for endpoints evaluating the change from week 0) or excluding timing will be used. The timing by quarters or halves is defined as too restrictive if the imputation model cannot be fit due to inadequate numbers of retrieved subjects in 1 or more groups. If the imputation model still cannot be fit after excluding timing then the model will be further reduced until the model can be fit.


31 March 2020 | Novo Nordisk 1.0 Final 14 of 24

Reduction will be done in a fixed order by first removing gender, then collapsing the two highest baseline BMI-groups into one (≥35) and finally removing baseline BMI-groups. If no LAO-OT exists post-baseline then the LAO-OT will be the baseline body weight and the timing will be the first interval. If any subjects are MT, an imputation model for missing body weight measurements at week 68 for MT subjects will also be defined using AT subjects in a similar way. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 68 body weight values for each randomised treatment arm. This will be done 1,000 times and results in 1,000 complete data sets.

- 2. Analysis: Analysis of each of the 1,000 complete data sets, using the analysis model (ANCOVA) results in 1,000 estimations.
- 3. **Pooling**: Integrates the 1,000 estimation results into a final result using Rubin's formula.

Based on NN9536-4153 phase 2 results 1,000 copies should be sufficient to establish stable results. If 1,000 copies are insufficient, 10,000 copies will be used. The multiple imputations will be generated using Novo Nordisk trial number 95364376 as seed number. In addition to the seed number, it is specified that the dataset is sorted by subject ID.

### Sensitivity analyses

Jump to reference multiple imputation approach (J2R-MI): Missing values of body weight at week 68 (MT and MD) for both the semaglutide 2.4 mg and semaglutide placebo group are imputed by sampling among all available assessments at week 68 in the semaglutide placebo group (AT and AD). This approach makes the assumption that subjects instantly after discontinuation lose any effect of randomised treatment beyond what can be expected from semaglutide placebo treatment as adjunct to reduced-calorie diet and increased physical activity. The multiple imputation approach is done as above with the first step replaced by

1. **Imputation**: Defines an imputation model using semaglutide placebo subjects from FAS with a week 68 measurement (AT and AD). The model will be a linear regression of body weight (kg) at week 68 with gender (male/female), BMI (kg/m<sup>2</sup>) (in categories 27-<35, 35-<40,  $\ge$ 40) as factors and baseline (randomisation) body weight (kg) as covariate. No interactions will be included. If the imputation model cannot be fit due to inadequate numbers of retrieved subjects in 1 or more groups, then the imputation model will be reduced until the model can be fit. Reduction will be done in a fixed order by first removing gender, then collapsing the two highest baseline BMI-groups into one ( $\geq$ 35) and finally removing baseline BMI-groups. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 68 body weight values for each randomised treatment arm. This will be done 1,000 times and results in 1,000 complete data sets.


31 March 2020 | Novo Nordisk 1.0 Final 15 of 24

The jump to reference approach is the basis for the sample size calculations.

A single imputation approach as done by Sacks<sup>4</sup> (S1-SI and S2-SI): Missing weight measurements at week 68 for non-retrieved subjects (MD) are imputed using a weight regain rate of 0.3 kg/month after LAO but truncated at no change from baseline whenever the extrapolation would lead to a positive weight gain relative to baseline. If a subject's weight at drug discontinuation represented a gain in weight relative to baseline, no additional gain will be imputed, and the unfavourable gain is carried forward to week 68. The weight regain imputation will be done for both randomised arms (S1-SI). Additionally, a version where only the semaglutide 2.4 mg arm uses the regain rate while the semaglutide placebo arm uses last available observation (corresponding to a weight regain rate of 0 kg/month) will be performed (S2-SI). For both versions, missing weight measurements at week 68 for subjects on randomised treatment (MT) are imputed by using LAO.

Tipping-point multiple imputation analysis (TP-MI): First, missing data are imputed according to the primary multiple imputation approach. Then, a penalty is added to the imputed values at week 68. The approach is to explore a range of penalties for both treatment groups, and the impact these would have on the study conclusions. The 2-dimensional space of penalties covering the range from -30% to 30% will be explored for both treatment groups. This sensitivity analysis evaluates the robustness of the superiority conclusions to departures from the observed change in body weight in both treatment groups.

Mixed model for repeated measurements (MMRM): This 'MMRM for effectiveness' will use all assessments regardless of adherence to randomised treatment, including assessments at week 68 for retrieved drop-outs (AD). The MMRM for effectiveness will be fitted using the same factor and covariate as for the primary analysis all nested within visit. An unstructured covariance matrix for measurements within the same subject will be employed, assuming that measurements for different subjects are independent.


31 March 2020 | Novo Nordisk 1.0 Final 16 of 24



Figure 2-1 Illustration of imputation approaches for the primary estimand


31 March 2020 | Novo Nordisk 1.0 Final 17 of 24

### Analysis addressing the secondary estimand

The secondary estimand for % weight change addresses the efficacy of semaglutide 2.4 mg and will be assessed using a 'MMRM for efficacy'. Week 68 assessments for retrieved drop-outs (AD) are not used in this analysis. The MMRM for efficacy will use assessments only from subjects who are taking the randomised treatment until end of treatment or until first discontinuing of randomised treatment. The derived date of the second consecutive missed dose will be used as the latest date for using assessments in this MMRM. The assessment closest in time and before the derived date of the second consecutive missed dose will be used as last assessment on randomised treatment. For subjects who initiate rescue interventions before completion or first discontinuing of randomised treatment, the date of starting weight management drugs or undergoing bariatric surgery will be used as latest date for using assessments in this MMRM. Similarly, the assessment closest in time and before the date of starting weight management drugs or undergoing bariatric surgery will be used as last assessment on randomised treatment. The MMRM for efficacy will be fitted using % weight change and the same factor and covariate as for the primary analysis all nested within visit. An unstructured covariance matrix for measurements within the same subject will be employed, assuming that measurements for different subjects are independent.

An overview of all analysis and imputation methods to address the primary and secondary estimands for the primary endpoint is given in Table 2-3.

#### 2.3.2 Secondary endpoints

#### 2.3.2.1 **Confirmatory secondary endpoints**

Confirmatory secondary endpoints are listed in Section 4.2.2.1 in the protocol and are all included in the fixed-sequence statistical strategy, see above. All tests are tests of superiority of semaglutide 2.4 mg to semaglutide placebo.

### Analyses addressing the primary estimand

All confirmatory secondary endpoints will be analysed using the same imputation approach as used for the primary endpoint and to address the primary estimand. The imputation model is the same as for the primary endpoint with body weight replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % weight change with baseline (randomisation) body weight replaced by the baseline (randomisation) assessment of the endpoint to be analysed.

### Analyses addressing the secondary estimand

The confirmatory secondary endpoints will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoint.

Sensitivity analyses for confirmatory secondary endpoints

For all continuous confirmatory secondary endpoints a sensitivity analysis using jump to reference as imputation approach will be carried out.

| Statistical Analysis Plan | Date: | 31 March 2020 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: 2017-003473-34 | Page: | 18 of 24 | |

An overview of all analysis and imputation methods to address the primary and secondary estimands for confirmatory secondary endpoints is given in <u>Table 2-3</u>.

Table 2-3 Analysis and imputation methods to address the primary and secondary estimands for the primary and confirmatory secondary endpoints in the statistical testing hierarchy

| Objective | Endpoint | Test | Endpoint | Estimand | Analysis | Statistical | Imputation | Sensitivity |
|---|---|---|---|---|---|---|---|---|
| | _ | order | type | | set | model | approach | analyses |
| Primary en | rimary endpoint | | | | | | | |
| From randor | misation (week 20) to week 6 | 8 | | | | | | |
| Primary | % weight change | 1 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI<br>S1-SI<br>S2-SI<br>TP-MI<br>MMRM |
| | | | | Secondary | FAS | MMRM | - | - |
| Confirmato | ry secondary endpoints | | | | | | | |
| From rando | misation (week 20) to week 6 | 8 | | | | | | |
| Primary | WC change (cm) | 2 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI |
| | | | | Secondary | FAS | MMRM | - | - |
| Secondary | sBP change (mmHg) | 3 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI |
| | | | | Secondary | FAS | MMRM | - | - |
| Secondary | SF-36 PF score change | 4 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI |
| | | | | Secondary | FAS | MMRM | - | - |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; J2R-MI = jump to reference multiple imputation; S1-SI and S2-SI = single imputation as done by Sacks; TP-MI = tipping point multiple imputation; MMRM = mixed model for repeated measurements; WC = waist circumference; sBP = systolic blood pressure; SF-36 = Short Form 36 v2.0 acute; PF = physical functioning;

Test order refers to the order of the endpoint in the statistical test hierarchy outlined in Table 2-2

### 2.3.2.2 Supportive secondary endpoints

Supportive secondary endpoints are listed in Section 4.2.2.2 in the protocol. All tests are tests of superiority of semaglutide 2.4 mg to semaglutide placebo.

### Analyses addressing the primary estimand

The effect-related supportive secondary endpoints will be analysed using the same imputation approach as used for the primary endpoint and to address the primary estimand. The imputation model is the same as for the primary endpoint with body weight replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % weight change with baseline (randomisation) body weight replaced by the baseline (randomisation) assessment of the endpoint to be analysed.

The statistical model for responder endpoints relating to clinical outcome assessments will be logistic regression with randomised treatment as a factor and the baseline (randomisation) assessment of the endpoint to be analysed as covariate.

The supportive secondary endpoint subjects who gain weight from randomisation (week 20) to week 68 (yes/no)' is used to describe weight maintenance. It will be analysed using logistic regression with randomised treatment as a factor and body weight (kg) at baseline (randomisation) as covariate.


31 March 2020 | Novo Nordisk 1.0 Final 19 of 24

For lipids and fasting serum insulin a multiplicative model will be used, i.e. the ratio between post randomisation measurements and baseline (randomisation) will be calculated instead of differences, and both the dependent variable and covariate will be log-transformed.

### Analyses addressing the secondary estimand

The supportive secondary endpoints will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoint.

The secondary estimand for weight gain responders will be assessed using the same MMRM for efficacy except that body weight (kg) will be used as response variable in the model. For subjects with missing body weight at week 68, individual values for body weight will be predicted from the MMRM and used to classify each subject as weight gain responder or not. This classification will then be analysed using a logistic regression model with randomised treatment as a factor and baseline (randomisation) body weight (kg) as covariate.

The secondary estimand for responder endpoints relating to clinical outcome assessments will be analysed using the same MMRM for efficacy as described for weight gain responders, where baseline (randomisation) body weight (kg) is replaced by baseline (randomisation) assessment of the endpoint to be analysed.

### Analyses addressing the tertiary estimand

The effect-related supportive secondary endpoints addressing the tertiary estimand will be analysed using the same imputation approach as used for the primary endpoint, where baseline (randomisation) body weight (kg) is replaced by baseline (week 0) body weight (kg). The continuous endpoint on body weight will be analysed using ANCOVA with factor and covariate as for the primary endpoint % weight change with the baseline (randomisation) value replaced with baseline (week 0). The binary endpoints on body weight will be analysed using logistic regression with randomised treatment as a factor and baseline (week 0) assessment of body weight as covariate.

### Analyses addressing the quaternary estimand

The effect-related supportive secondary endpoints addressing the quaternary estimand will be analysed using the same MMRM for efficacy described for the primary endpoint, where baseline (randomisation) body weight (kg) is replaced by baseline (week 0) body weight (kg).

The quarternary estimand for bw responders will be assessed using the same MMRM for efficacy described for the secondary estimand for the weight gain responders, where baseline (randomisation) body weight (kg) is replaced by baseline (week 0) body weight (kg).

*Sensitivity analyses for supportive secondary endpoints* 

For supportive secondary endpoints no sensitivity analysis will be carried out.


31 March 2020 | Novo Nordisk 1.0 Final 20 of 24

### Additional considerations for statistical analyses

To evaluate the predictive value of short-term weight changes for long-term benefit of the use of semaglutide 2.4 mg, subjects will be categorised based on the weight change achieved in the run-in phase. If the weight change from week 0 to week 20 exceeds a certain pre-specified threshold subjects are classified as early "responders" whereas subjects are classified as early "nonresponders" if the weight has changed less than the pre-specified threshold. Different thresholds of 3%, 4% and 5% will be investigated. These sub-group analyses will be done using the primary endpoint and the statistical model described for the primary endpoint. These analyses will be presented in a report separate from the Clinical Trial Report.

#### **Analysis of safety endpoints**

The safety endpoint pulse from randomisation (week 20) to week 68 will be analysed using an MMRM for efficacy as described in Section 2.3.1. For pulse from week 0 to randomisation (week 20), amylase, lipase and calcitonin descriptive statistics will be provided. The analysis of calcitonin will be stratified by gender.

Adverse events will be defined as "treatment-emergent" (TEAE), if the onset of the event occurs in the on-treatment period (see definition in Section 2.2). TEAEs and SAEs will be summarised by descriptive statistics, such as frequencies and rates. No formal statistical inference will be carried out based on the number of TEAEs and SAEs. All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA).

An overview of all analysis and imputation methods to address the primary, secondary, tertiary and quaternary estimands for supportive secondary endpoints is given in Table 2-4.


 Date:
 31 March 2020

 Version:
 1.0

 Status:
 Final

 Page:

Table 2-4 Analysis and imputation methods to address the primary, secondary, tertiary and quaternary estimands for supportive secondary endpoints

| Objective | Endpoint | Endpoint<br>type | Estimand | Analysis<br>set | Statistical model | Imputation approach | Sensitivity analyses |
|---|---|---|---|---|---|---|---|
| Supportive s | secondary endpoints (effect related) | | | | • | | |
| | misation (week 20) to week 68 | | | | | | |
| Primary | Weight change (kg) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| 3 | | | Secondary | FAS | MMRM | - | - |
| Primary | BMI change (kg/m <sup>2</sup> ) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| , | | | Secondary | FAS | MMRM | - | - |
| Secondary | HbA <sub>1c</sub> change (%, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| , | | | Secondary | FAS | MMRM | - | |
| Secondary | FPG change (mg/dL,mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| , | | | Secondary | FAS | MMRM | - | |
| Secondary | Fasting serum insulin change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| , | (mIU/L, pmol/mol) | | Secondary | FAS | MMRM | - | |
| Secondary | dBP change (mmHg) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| , | | | Secondary | FAS | MMRM | - | |
| Secondary | Total cholesterol change (mg/dL, | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | mmol/mol) | | Secondary | FAS | MMRM | - | |
| Secondary | HDL change (mg/dL, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| Secondary | ing united in the state of the | Commuous | Secondary | FAS | MMRM | - | |
| Secondary | LDL change (mg/dL, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| Secondary | LDE change (mg/aE, mmor/mor) | Continuous | Secondary | FAS | MMRM | - | |
| Secondary | VLDL change (mg/dL, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| Secondary | VEDE change (mg/dE, mmor/mor) | Continuous | Secondary | FAS | MMRM | KD-WII | _ |
| Secondary | FFA change (mg/dL, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| Secondar y | TTA change (mg/dL, mmol/mor) | Continuous | Secondary | FAS | MMRM | KD-WII | - |
| Secondary | Triglycerides change (mg/dL, | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| Secondar y | mmol/mol) | Continuous | Secondary | FAS | MMRM | KD-WII | - |
| Secondary | SF-36 PF score responders # | Binary | Primary | FAS | LR | RD-MI | _ |
| Secondary | Sr-30 FF score responders # | Billary | Secondary | FAS | LR | MMRM | - |
| Secondary | SF-36 RP score change | Continuous | Primary | FAS | ANCOVA | RD-MI | |
| Secondary | SF-36 KP score change | Continuous | | FAS | MMRM | KD-MI | - |
| C 1 | SF-36 BP score change | Continue | Secondary<br>Primary | | | - DD M | |
| Secondary | SF-36 BP score change | Continuous | | FAS | ANCOVA | RD-MI | - |
| G 1 | OF 24 CH | a ii | Secondary | FAS | MMRM | - DD 14 | |
| Secondary | SF-36 GH score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| 0 1 | OF 26 MT | a ii | Secondary | FAS | MMRM | -<br>DD 14 | |
| Secondary | SF-36 VT score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| o . | gracer . | a ii | Secondary | FAS | MMRM | - | |
| Secondary | SF-36 SF score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | |
| Secondary | SF-36 RE score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | |
| Secondary | SF-36 MH score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | |
| Secondary | SF-36 PCS score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | |
| Secondary | SF-36 MCS score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | |
| Primary | Proportion of subjects who gain | Binary | Primary | FAS | LR | RD-MI | - |
| - | weight (%) | | Secondary | FAS | LR | MMRM | |

Statistical Analysis Plan

Date: 31 March 2020 Novo Nordisk

 Trial ID: NN9536-4376
 Version:
 1.0

 UTN: U1111-1201-0898
 Status:
 Final

 EudraCT No.: 2017-003473-34
 Page:

| From week ( | to week 68 | | | | | | |
|---|---|---|---|---|---|---|---|
| Secondary | % weight change | Continuous | Tertiary | FAS | ANCOVA | RD-MI | - |
| | | | Quarternary | FAS | MMRM | - | |
| Secondary | Weight reduction <0% | Binary | Tertiary | FAS | LR | RD-MI | - |
| | | | Quarternary | FAS | LR | MMRM | |
| Secondary | Weight reduction ≥5% | Binary | Tertiary | FAS | LR | RD-MI | - |
| | | | Quarternary | FAS | LR | MMRM | |
| Secondary | Weight reduction ≥10% | Binary | Tertiary | FAS | LR | RD-MI | - |
| | | | Quarternary | FAS | LR | MMRM | |
| Secondary | Weight reduction ≥15% | Binary | Tertiary | FAS | LR | RD-MI | - |
| | | | Quarternary | FAS | LR | MMRM | |
| Secondary | Weight reduction ≥20% | Binary | Tertiary | FAS | LR | RD-MI | - |
| | | | Quarternary | FAS | LR | MMRM | |
| Supportive | secondary endpoints (safety relat | ed) | | | | | |
| From week ( | to randomisation (week 20) | | | | | | |
| Secondary | Number of TEAEs | Continuous | - | SAS | - | - | - |
| Secondary | Number of SAEs | Continuous | - | SAS | - | - | - |
| Secondary | Pulse change (bpm) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Amylase change (U/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Lipase change (U/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Calcitonin change (ng/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| From rando | nisation (week 20) to week 68 / 75 | • | • | | • | • | • |
| Secondary | Number of TEAEs | Continuous | - | SAS | - | - | - |
| Secondary | Number of SAEs | Continuous | - | SAS | - | - | - |
| Secondary | Pulse change (bpm) | Continuous | - | SAS | MMRM | - | - |
| Secondary | Amylase change (U/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Lipase change (U/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Calcitonin change (ng/L) | Continuous | - | SAS | Descriptive statistics | - | - |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; MMRM = mixed model for repeated measurements; BMI = body mass index; HbA1c = Hemoglobin A1c; FPG = fasting plasma glucose; dBP = diastolic blood pressure; HDL = high density lipoprotein; LDL = low density lipoprotein; VLDL = very low density lipoprotein; FFA = free fatty acids; LR = logistic regression; SF-36 = Short Form 36 v2.0 acute; PF= Physical Functioning; RP = Role-Physical; BP = Bodily Pain; GH = General Health; VT = Vitality; SF = Social Functioning; RE = Role-Emotional; MH = Mental Health; PCS = Physical component summary; MCS = Mental component summary; TEAEs = treatment emergent adverse events; SAEs = serious adverse events; # responder value = 4.3

### 2.3.3 Exploratory endpoints

Exploratory endpoints are listed in Section 4.2.3 in the protocol. Observed data for exploratory endpoints will be summarised by descriptive statistics.

### 2.3.4 Other analyses

All collected data that were not defined as endpoints will be summarised by descriptive statistics.

#### 2.4 Pharmacokinetic and/or pharmacodynamic modelling

Not applicable for this trial.


31 March 2020 | Novo Nordisk 1.0 Final 23 of 24

#### 3 Changes to the statistical analyses planned in the protocol

The main analyses were described in the protocol for the trial NN9536-4376. However, clarifications and more detailed descriptions of endpoints and analyses are provided in this SAP. The changes from the protocol of NN9536-4376 are summarised below:

#### 3.1 Trial specific changes

- Ouaternary estimand has been defined to account for analyses based on the hypothetical estimand for weight related endpoints from week 0 to week 68.
- Description of the MMRM for efficacy for weight gain responders has been added.
- It has been clarified that the safety endpoint pulse from week 0 to randomisation (week 20) will not be analysed but reported with descriptive statistics.
- It has been clarified that the "early responder" analyses will not be presented in the Clinical Trial Report, but in a separate report.

#### 3.2 **Changes applied across STEP trials**

- The supportive secondary endpoint "Body weight reduction ≥ 20% from baseline at week 0" was added.
- It was clarified that subjects in the FAS/SAS will be evaluated "as randomised"/"as treated".
- In the text describing that "In general, the on-treatment period will therefore be from the date of first trial product administration to date of last trial product administration" the following has been added "(+14 days)" to emphasize that the lag-time after last trial product administration is included in the on-treatment period.
- All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA).
- The text explaining how to handle missing baseline values has been changed to make it clear that if no eligible observation at or before randomisation is available then the mean of baseline values across all subjects is used as baseline value.
- It is clarified that RD-MI imputation is performed according to the timing of last available observation during the on-treatment period (LAO-OT). This is true for all endpoints. This is to clarify that the grouping of subjects according to timing is as in McEvoy<sup>2</sup>. Furthermore it is clarified that the LAO-OT must be prior to the landmark visit (week 68)
- BMI group "27-<35" in the RD-MI imputation has been updated to "\( \sigma 35\)" to reflect that some subjects loose weight between screening and randomisation and therefore can have a BMI  $\leq$  27 kg/m $^{\circ}$ 2 at the randomisation visit.
- In grouping of retrieved subjects by timing of LAO-OT in the RD-MI procedure, it is clarified that timing by quarters or halves is defined as too restrictive if the imputation model cannot be fit due to inadequate numbers of retrieved subjects in 1 or more groups. Furthermore it is described how a model reduction will be performed if needed.


 Date:
 31 March 2020
 Novo Nordisk

 Version:
 1.0

 Status:
 Final

 Page:

• It is clarified that if no post-baseline LAO-OT exist, then LAO-OT will be the baseline value and the timing of LAO-OT will be the first interval.

- In all multiple imputation procedures, in addition to the seed number, it is specified that the dataset is sorted by subject ID.
- The TP-MI procedure has been updated to be a 2-way tipping point analysis in which penalties are applied to both treatment groups (semaglutide 2.4 mg and placebo).
  - The rational for the changed TP-MI procedure is as follows: "To confirm the robustness of superiority conclusions using a tipping point analysis, we believe that a 2-way tipping point analysis represents the real-world situation for missing data from the both treatment arms (semaglutide and placebo). We would like to see departures from the treatment difference by varying both treatment arms rather than only adding a penalty to the active treatment arm (semaglutide). Additionally, please include interpretations for the varying scenarios and how likely they would be seen in a real-world setting." (from FDA response letter 17 May 2018).
- It is specified that fasting serum insulin will be log-transformed and analysed using a multiplicative model.
- It is specified that lipids, FPG and fasting serum insulin will also be analysed in SI-units.
- Text and tables have been updated to reflect that analyses for all non-weight related endpoints based on the secondary estimand and analyses for all weight related endpoints based on the quaternary estimand are to be done.

## 4 References

- 1. International Conference on Harmonisation. ICH Harmonised Tripartite Guideline. Topic E10: Choice of control group and related issues in clinical trials, 20 July 2000.
- 2. McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6.
- 3. Carpenter JR, Roger JH, Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat. 2013;23(6):1352-71.
- 4. Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, et al. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009;360(9):859-73.

Semaglutide s.c. 2.4 mg once weekly Trial ID: NN9536-4376 (STEP 4) Clinical Trial Report MedDRA searches


17 April 2020 | Novo Nordisk 1.0 Final 1 of 7

# **Clinical Trial Report**

Trial ID: NN9536-4376 (STEP 4)

MedDRA searches within safety focus areas

### CONFIDENTIAL


17 April 2020 | Novo Nordisk 1.0 Final 2 of 7

# **Table of contents**

| | | Page |
|-----|----------------------------------------------------------|------|
| Tal | ble of contents | 2 |
| Lis | et of abbreviations and definitions of terms | 3 |
| 1 | MedDRA searches for safety focus areas in project NN9536 | 4 |
| 2 | Abuse and misuse | 4 |
| 3 | Acute renal failure | 4 |
| 4 | Allergic reactions | 4 |
| 5 | Cardiovascular disorders | 4 |
| 6 | Drug-related hepatic disorders | 5 |
| 7 | Gallbladder-related disorders | 5 |
| 8 | Gastrointestinal disorders | 5 |
| 9 | Hypoglycaemia | 5 |
| 10 | Injection site reactions | 5 |
| 11 | Malignant tumours | 6 |
| 12 | Medication errors | 6 |
| 13 | Neoplasms | 6 |
| 14 | Overdose | 6 |
| 15 | Pancreatitis | 7 |
| 16 | Psychiatric disorders | 7 |
| 17 | Rare events | 7 |

Semaglutide s.c. 2.4 mg once weekly Trial ID: NN9536-4376 (STEP 4) Clinical Trial Report MedDRA searches


17 April 2020 | Novo Nordisk 1.0 Final 3 of 7

# List of abbreviations and definitions of terms

ΑE adverse event HLT high level term

MedDRA Medical Dictionary for Regulatory Activities

NEC not elsewhere classified

Novo Nordisk MedDRA query NNMQ

PT preferred term

**SMQ** standardised MedDRA query

SOC system organ class Semaglutide s.c. 2.4 mg once weekly Trial ID: NN9536-4376 (STEP 4) Clinical Trial Report MedDRA searches


17 April 2020 | Novo Nordisk Final 4 of 7

#### MedDRA searches for safety focus areas in project NN9536 1

The MedDRA search strings in this document (ordered alphabetically) were used for the NN9536 submission documents. The same search strings were used for the STEP 1-4 clinical trial reports. The MedDRA version used was 22.1.

#### 2 Abuse and misuse

Custom query (NNMQ Abuse and Misuse):

- SMQ Drug abuse and dependence, narrow terms only
- HLT Intentional product misuses
- Additional PTs:
  - Poisoning deliberate
  - Intentional dose omission
  - o Performance enhancing product use
  - Completed suicide
  - o Intentional self-injury
  - Suicide attempt
  - Assisted suicide
  - Suspected suicide attempt
  - Suspected suicide.

#### 3 Acute renal failure

SMQ Acute renal failure, narrow terms only

#### 4 Allergic reactions

Custom Query (NNMQ Allergic reactions) – only narrow terms from the following:

- SMQ Anaphylactic reaction
- SMQ Angioedema
- SMQ Severe cutaneous adverse reactions
- SMQ Anaphylactic/anaphylactoid shock conditions
- SMQ Hypersensitivity

#### Cardiovascular disorders 5

Custom query (NNMQ Cardiovascular disorders). Broad and narrow terms from the following:

- SMQ Central nervous system vascular disorders
- **SMQ Vasculitis**

Semaglutide s.c. 2.4 mg once weekly
Trial ID: NN9536-4376 (STEP 4)
Clinical Trial Report
MedDRA searches

Date: 17 April 2020 Version: 1.0
Status: Final
Page: 5 of 7

- SMQ Ischaemic heart disease
- SMQ Cardiac arrhythmias
- SMQ Cardiac failure
- SMQ Cardiomyopathy
- SMQ Embolic and thrombotic events
- SMQ Shock
- SMQ Torsade de pointes/QT prolongation

# 6 Drug-related hepatic disorders

SMQ Drug related hepatic disorders - comprehensive search

## 7 Gallbladder-related disorders

Custom query (NNMQ Gallbladder-related disorders). Narrow terms from the following:

- SMQ Functional, inflammatory and gallstone related biliary disorders
- SMQ Infectious biliary disorders

## 8 Gastrointestinal disorders

Custom query (NNMQ Gastrointestinal disorders SOC):

• SOC Gastrointestinal disorders, primary terms only

# 9 Hypoglycaemia

SMQ Hypoglycaemia, narrow terms only

# 10 Injection site reactions

Custom query (NNMQ Injection site reactions), both primary and secondary terms from the following:

- HLT Administration site reactions NEC
- HLT Application and instillation site reactions
- HLT Infusion site reactions
- HLT Injection site reactions

Semaglutide s.c. 2.4 mg once weekly Trial ID: NN9536-4376 (STEP 4) Clinical Trial Report MedDRA searches


17 April 2020 | Novo Nordisk 1.0 Final 6 of 7

# **Malignant tumours**

SMQ Malignant tumours

# 12 Medication errors

SMQ Medication errors.

# 13 Neoplasms

Custom query (NNMQ Neoplasms)

- SOC Neoplasms benign, malignant and unspecified (incl cysts and polyps), primary and secondary terms
- SMQ Biliary neoplasms
- SMQ Breast neoplasms, malignant and unspecified
- SMQ Liver neoplasms, benign (incl cysts and polyps)
- SMQ Liver neoplasms, malignant and unspecified
- SMQ Malignancies
- SMQ Malignant lymphomas
- SMQ Oropharyngeal neoplasms
- SMQ Ovarian neoplasms, malignant and unspecified
- SMQ Premalignant disorders
- SMQ Prostate neoplasms, malignant and unspecified
- SMQ Skin neoplasms, malignant and unspecified
- SMQ Uterine and fallopian tube neoplasms, malignant and unspecified

## 14 Overdose

Custom query (NNMQ Overdose):

- **HLT Overdoses NEC**
- Additional PTs:
  - Accidental overdose
  - o Completed suicide
  - Suicide attempt
  - Suspected suicide attempt
  - Suspected suicide

| Semaglutide s.c. 2.4 mg once weekly Trial ID: NN9536-4376 (STEP 4) Clinical Trial Report MedDRA searches | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 17 April 2020 <b>Novo Nord</b> 1.0 Final 7 of 7 | lisk |
|---|---|---|---|---|
|---|---|---|---|---|

### 15 Pancreatitis

Custom query (NNMQ Pancreatitis), narrow terms from the following:

- SMQ Acute pancreatitis
- HLT Acute and chronic pancreatitis, primary and secondary terms

# 16 Psychiatric disorders

Custom query:

• SOC Psychiatric disorders, primary terms only

## 17 Rare events

Custom query (NNMQ Rare events) excluding events that are included in other safety focus areas:

- SMQ Agranulocytosis, narrow terms only
- SMQ Guillain-Barre syndrome, narrow terms only
- SMQ Haematopoietic cytopenias affecting more than one type of blood cell, broad and narrow terms
- SMQ Haematopoietic leukopenia, broad and narrow terms
- SMQ Haematopoietic thrombocytopenia, narrow terms only
- SMQ Interstitial lung disease, narrow terms only
- SMQ Neuroleptic malignant syndrome, narrow terms only
- SMQ Pseudomembranous colitis, narrow terms only
- SMQ Retroperitoneal fibrosis, narrow terms only
- SOC Congenital, familial and genetic disorders, (all terms are primary PTs)
- HLT Angioedemas, primary and secondary routed PTs
- HLT Glomerulonephritis and nephrotic syndrome, primary and secondary routed PTs
- HLT Nephritis NEC, primary and secondary routed PTs
- Additional PTs:
  - o Disseminated intravascular coagulation
  - o Hepatic lymphocytic infiltration
  - o Multiple organ dysfunction syndrome